CLINICAL TRIAL: NCT01685957
Title: Optimal Dietary Treatment of Obese Adults
Acronym: OPDIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitalsenheden Vest (Other)
Responsible Party: Principal Investigator, Allan Stubbe Christensen, MHSc, RD, Hospitalsenheden Vest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASC-01-2012
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Overweight
Keywords: Weight loss; Dietary intervention; Self-help book; Cooking; Dietitian; Dietary therapy
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard dietary treatment (STD) (Active Comparator): Dietary treatment - 6 individual sessions with a registered dietitian
  Interventions: Behavioral: Standard dietary treatment (STD)
- "Ned i vaegt" (NIV) (Experimental): Dietary treatment - 3 individual sessions and 3 group sessions. All sessions with a registered dietitian.
  Interventions: Behavioral: "Ned i vaegt" (NIV)
- "Verdens bedste kur" (VBK) (Experimental): Dietary treatment - 3 individual sessions and 3 group sessions. All sessions with a registered dietitian.
  Interventions: Behavioral: "Verdens bedste kur" (VBK)

INTERVENTIONS:
Behavioral: Standard dietary treatment (STD) — This group will receive 6 one-on-one sessions with a registered dietitian. Total time spent is 6½ hour. Dietary treatment is based national guidelines and counseling is individualized and tailored to the patient's needs and goals.
  Arms: Standard dietary treatment (STD)
Behavioral: "Ned i vaegt" (NIV) — This group will receive 3 individual sessions and 3 group sessions. All sessions are with a registered dietitian. Total time spent is 15½ hour. The group sessions consist of 1 hour theory and 2½ hour cooking skills. The whole intervention is based on a danish self-help weightloss book which is based on the national dietary guidelines. Focus is to learn to make "normal" danish dishes in a more healthy way both ingredients, cooking, composition and quantity. They also learn about changing habits, making realistic goals and using their motivation.
  Arms: "Ned i vaegt" (NIV)
Behavioral: "Verdens bedste kur" (VBK) — This group will receive 3 individual sessions and 3 group sessions. All sessions are with a registered dietitian. Total time spent is 15½ hour. The group sessions consist of 1 hour theory and 2½ hour cooking skills. The whole intervention is based on a danish self-help weightloss book which is based on "new nordic diet" and are a relative low-GI and high-protein diet. Focus is to learn to make new healthy dishes both ingredients, cooking and composition. They also learn about making realistic goals.
  Arms: "Verdens bedste kur" (VBK)

SUMMARY:
Recent decades have shown an alarming increase in obesity. Obesity is associated with high costs for both the individual and for society. It is therefore important to prevent and treat obesity. The investigators believe that if you add a self-help weightloss book and teach cooking skills to a standard dietary treatment, then it will result in greater weight loss than with dietary treatment alone. However, this has not yet been studied. Since it will require more resources, it is important to investigate whether it also works better before changing the current treatment.

Hypothesis: Conventional dietary treatment supplemented with a self-help weightloss book and cooking classes are more effective than dietary treatment alone in changes in body weight and body composition in obese persons over a period of 12 months. There is no difference if the intervention are based on the national dietary guidelines or a relative low-gi and high-protein diet.

Secondary to investigate the impact the interventions have; on diet quality and quantity, on markers of metabolic syndrome and on how many subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25
* Waist: female ≥ 88 cm; male ≥ 102 cm)
* Stable weight for the past three month (+- 5 kilogram)
* Motivated to make changes in their dietary habits

Exclusion Criteria:

* Waist > 150 cm
* Significant cardiovascular, renal or endocrine disease
* Psychiatric history
* Treatment with steroids
* Alcohol- or drug-addiction
* Pregnancy or lactation
* Obesity surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Body weight | From week 0 to week 52

SECONDARY OUTCOMES:
Blood pressure | From week 0 to week 52
  Both systolic and diastolic blood pressure
Dexa-scan (body composition) | From week 0 to week 52
Waist circumference | From week 0 to week 52
Biomarkers in blood samples | From week 0 to week 52
  Lipid profile (total-cholesterol, LDL, HDL, triglyceride), fasting-glucose, HbA1c
Quality of life | From week 0 to week 52
  EQ-5D-5L
Dietary intake | From week 0 to week 52
  Diet records

CONTACTS AND LOCATIONS:
Overall Officials: Allan S Christensen, MHSc, Principal Investigator — Department of Nutrition, Regional Hospital West Jutland, Denmark; Lone Viggers, MSc, Principal Investigator — Department of Nutrition, Regional Hospital West Jutland, Denmark
Locations (1):
- Department of Nutrition, Regional Hospital West Jutland, Denmark, Holstebro, Denmark